CLINICAL TRIAL: NCT02227147
Title: An 8-week Phase II, Multicenter, Randomized, Double-masked, Vehicle Controlled Parallel Group Study With a 24 or 32 Week Follow-up to Evaluate the Efficacy of rhNGF 20 µg/ml vs Vehicle in Patients With Stage 2 and 3 Neurotrophic Keratitis
Brief Title: Evaluation of Efficacy of 20 µg/ml rhNGF New Formulation (With Anti-oxidant) in Patients With Stage 2 and 3 NK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0214
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Neurotrophic Keratitis
Keywords: Neurotrophic Keratitis
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhNGF 20 µg/ml (Experimental): rhNGF 20 µg/ml eye drops solution, formulation containing anti-oxidant
  Interventions: Drug: rhNGF 20µg/ml
- Placebo (Placebo Comparator): Vehicle: formulation containing anti-oxidant
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: rhNGF 20µg/ml
  Other Names: cenegermin
  Arms: rhNGF 20 µg/ml
Other: Placebo — Formulation containing antioxidant
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 20 µg/ml 6 times a day of rhNGF eye drops solution (formulation containing anti-oxidant) compared to vehicle (formulation containing anti-oxidant) given 6 times a day. The evaluation of efficacy is intended as:

* complete healing of stage 2 (persistent epithelial defect) and 3 (corneal ulcer) neurotrophic keratitis (NK) as measured by the central reading center using corneal fluorescein staining,
* assessing the duration of complete healing,
* improvement in visual acuity and improvement in corneal sensitivity.

DETAILED DESCRIPTION:
An 8-week phase II, multicenter, randomized, double-masked, vehicle-controlled, parallel group study with a 24 or 32 week follow-up period to evaluate the efficacy of a formulation containing anti-oxidant of recombinant human nerve growth factor (rhNGF) in 20 μg/ml, eye drops solution versus vehicle containing anti-oxidant in patients with Stage 2 and 3 Neurotrophic Keratitis. The primary objective was to evaluate the efficacy of 20 μg/ml 6 times a day of recombinant human nerve growth factor (rhNGF) containing anti-oxidant, eye drops solution compared to vehicle (formulation containing anti-oxidant) given 6 times a day in inducing a complete healing of stage 2 (PED) and 3 (corneal ulcer) NK as measured by the central reading center, evaluating the clinical pictures of corneal fluorescein staining.

Secondary objectives were to assess the duration of complete healing, improvement in visual acuity and improvement in corneal sensitivity, and percentage of patients achieving complete corneal clearing defined as complete absence of staining on the modified Oxford Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients with stage 2 (persistent epithelial defect, PED) or stage 3 (corneal ulcer) neurotrophic keratitis (NK).
* PED or corneal ulceration of at least 2 weeks duration refractory to one or more conventional non-surgical treatments for neurotrophic keratitis.
* Evidence of decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant.
* Best corrected distance visual acuity (BCDVA) score ≤ 75 ETDRS (Early Treatment Diabetic Retinopathy Study)letters, (≥ 0.2 LogMAR, ≤ 20/32 Snellen or ≤ 0.625 decimal fraction) in the affected eye(s).
* No objective clinical evidence of improvement in the PED or corneal ulceration within the 2 weeks prior to study enrolment.
* Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the IRB (Institutional Review Board) for the current study.
* Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

* Any active ocular infection or active ocular inflammation not related to NK in the affected eye(s).
* Any other ocular disease requiring topical ocular treatment during the course of the study treatment period. No topical treatments other than the study medications provided by the study sponsor and allowed by the study protocol can be administered in the affected eye(s) during the course of the study treatment periods.
* Patients with severe vision loss with no potential for visual improvement in the opinion of the investigator as a result of the study treatment.
* Schirmer test without anesthesia ≤3 mm/5 minutes.
* Patients with severe blepharitis and/or severe meibomian gland disease.
* History of any ocular surgery (including laser or refractive surgical procedures) within the three months before study enrolment. (An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the stage 2 or 3 NK). Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period.
* Prior surgical procedure(s) for the treatment of NK with the exception of amniotic membrane transplantation. Patients previously treated with amniotic membrane transplantation may only be enrolled two weeks after the membrane has disappeared within the area of the PED or corneal ulcer or at least six weeks after the date of the amniotic membrane transplantation procedure.
* Patients previously treated with Botox injections used to induce pharmacologic blepharoptosis are eligible for enrolment only if the last injection was given at least 90 days prior to enrolment in the study.
* Anticipated need to use therapeutic contact lenses or contact lens wear for refractive correction during the study treatment period in the eye(s) with NK.
* Anticipated need for punctual occlusion during the study treatment period. Patients with punctual occlusion or punctual plugs inserted prior to the study are eligible for enrolment provided that the punctual occlusion is maintained during the study.
* Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting or perforation.
* Presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct.
* Any need for or anticipated change in the dose of systemic medications known to impair the function of the trigeminal nerve. These treatments are allowed during the study if initiated prior study enrolment provided they remain stable throughout the course of the study treatment periods.
* Known hypersensitivity to one of the components of the study or procedural medications (e.g. fluorescein).
* History of drug, medication or alcohol abuse or addiction.
* Use of any investigational agent within 4 weeks of screening visit.
* Participation in another clinical study at the same time as the present study.
* Females of childbearing potential are excluded from participation in the study if they meet any one of the following conditions: are currently pregnant or, have a positive result on the urine pregnancy test at the Randomization Visit or, intend to become pregnant during the study treatment period or, are breast-feeding or are not willing to use highly effective birth control measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Director — Dompé farmaceutici S.p.A., Milan
Locations (12):
- United States (12):
  - Loma Linda University Ophthalmology, Loma Linda, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Shiley Eye Center University of California, San Diego, California
  - Bascom Palmer Eye Institute University of Miami, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts Eye & Ear Infirmary, Boston, Massachusetts
  - Massachusetts Eye Research and Surgery Institution, Cambridge, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York Eye and Ear Infirmary, New York, New York
  - Penn Eye Care Scheie Eye Institute, Philadelphia, Pennsylvania
  - UPMC eye center, department of ophthalmology, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was competitive among the study sites, until the planned number of patients were randomized.
  Competitive recruitment was chosen to increase the speed of recruitment and to account for any difference in enrolment rate among study sites.
Groups:
- rhNGF 20 µg/ml: rhNGF 20 µg/ml eye drops solution, formulation containing anti-oxidant
  rhNGF 20µg/ml
- Vehicle: vehicle, formulation containing anti-oxidant
  Placebo Vehicle
Period: Controlled Treatment Period
Arm/Group | rhNGF 20 µg/ml | Vehicle
Started | 24 | 24
Completed | 18 | 21
Not Completed | 6 | 3
Not completed — Adverse Event | 4 | 3
Not completed — Other | 2 | 0
Period: Follow-up Period
Arm/Group | rhNGF 20 µg/ml | Vehicle
Started | 18 | 21
Completed | 15 | 16
Not Completed | 3 | 5
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 20 µg/ml | Vehicle | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 13 | 24
  >=65 years | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (13.85) | 54.5 (14.15) | 65.2 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Complete Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer Defined by Central Reviewer
Description: Percentage of patients achieving complete healing of the PED or corneal ulcer determined by corneal fluorescein staining at 8 weeks as defined by the central reading center on clinical pictures.
Time Frame: Week 8
Population: ITT population, LOCF. One patient (randomized to rhNGF although not eligible) had no post-baseline data, was assumed to be missing, and was excluded from the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 23 | 24
percentage of participants
  Completely healed | 70 | 29
  Not completely healed | 30 | 71
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Vehicle; Test type: Superiority; p = 0.006, Chi-squared; Difference in percentage = 40.4, 90.00% CI 2-sided [14.2 to 66.6]

2. Secondary Outcome: Complete Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer Defined by the Investigator
Description: Percentage of patients experiencing complete healing of the PED or corneal ulcer determined by corneal fluorescein staining at 8 weeks as measured by the investigator.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | rhNGF 20 µg/ml | Vehicle
Number analyzed (Participants) | 23 | 24
percentage of participants
  Completely healed | 65 | 29
  Not completely healed | 35 | 71
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Vehicle; Test type: Superiority; p = 0.013, Chi-squared; Difference in percentage = 36.1, 95.0% CI 2-sided [9.4 to 62.7]

3. Secondary Outcome: Complete Healing of the Persistent Epithelial Defect (PED) or Corneal Ulcer Defined by Central Reading Center and Investigator.
Description: Percentage of patients experiencing complete healing of the PED or corneal ulcer at 4, and 6 weeks as measured by the central reading center evaluating the clinical pictures and investigator.
Time Frame: At weeks 4 and 6
Population: LOCF, ITT population. One patient (randomized to rhNGF although not eligible) had no post-baseline data, was assumed to be missing, and was excluded from the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 23 | 24
percentage of participants
  Week 4 - central reviewer - yes | 56 | 38
  Week 4 - central reviewer - no | 44 | 62
  Week 6 - central reviewer - yes | 56 | 46
  Week 6 - central reviewer - no | 44 | 54
  Week 4 - investigator - yes | 56 | 42
  Week 4 - investigator - no | 44 | 58
  Week 6 - investigator - yes | 65 | 42
  Week 6 - investigator - no | 35 | 58
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; week 4 - central reviewer; Test type: Superiority; p = 0.191, Chi-squared; difference in percentage = 19.0, 95% CI 2-sided [-9.0 to 47.1]
Statistical Analysis 2: Comparison: rhNGF 20 µg/ml vs Placebo; week 6 - central reviewer; Test type: Superiority; p = 0.464, Chi-squared; difference in percentage = 10.7, 95% CI 2-sided [-17.7 to 39.1]
Statistical Analysis 3: Comparison: rhNGF 20 µg/ml vs Placebo; week 4 - investigator; Test type: Superiority; p = 0.308, Chi-squared; difference in percentage = 14.9, 95% CI 2-sided [-13.4 to 43.1]
Statistical Analysis 4: Comparison: rhNGF 20 µg/ml vs Placebo; week 6 - investigator; Test type: Superiority; p = 0.106, Chi-squared; difference in percentage = 23.6, 95% CI 2-sided [-4.2 to 51.3]

4. Secondary Outcome: Percentage of Patients With Complete Corneal Clearing
Description: Percentage of patients with complete corneal clearing at weeks 4, 6, and 8 defined as grade 0 on the modified Oxford scale. Grade 0 indicates the absence of conjunctival staining; grade V indicates severe conjunctival staining.
Time Frame: at weeks 4, 6, and 8
Population: LOCF, ITT population. Two patients (randomized to rhNGF although not eligible) had no post-baseline data, were assumed to be missing, and were excluded from the analyses.
Measure: Number; unit: percentage of participants
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 22 | 24
percentage of participants
  Week 4 - yes | 14 | 4
  Week 4 - no | 86 | 96
  Week 6 - yes | 9 | 8
  Week 6 - no | 91 | 92
  Week 8 - yes | 23 | 4
  Week 8 - no | 77 | 96
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; week 4; Test type: Superiority; p = 0.255, Chi-squared; difference in percentage = 9.5, 95% CI 2-sided [-6.9 to 25.9]
Statistical Analysis 2: Comparison: rhNGF 20 µg/ml vs Placebo; week 6; Test type: Superiority; p = 0.927, Chi-squared; difference in percentage = 0.8, 95% CI 2-sided [-15.6 to 17.1]
Statistical Analysis 3: Comparison: rhNGF 20 µg/ml vs Placebo; week 8; Test type: Superiority; p = 0.062, Chi-squared; difference in percentage = 18.6, 95% CI 2-sided [-0.7 to 37.8]

5. Secondary Outcome: Mean Change From Baseline in Best Corrected Distance Visual Acuity (BCDVA)
Description: Change in Best Corrected Distance Visual Acuity (BCDVA) from baseline to Week 8.
  Best Corrected Distance Visual Acuity consists of letters read at 4m only.
Time Frame: Baseline, Week 8
Population: LOCF, ITT Population
Measure: Mean (Standard Deviation); unit: letters read correctly
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 23 | 24
letters read correctly | 4.48 (9.25) | 4.33 (10.399)
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; Test type: Superiority; p = 0.745, ANCOVA; difference in least square means = 1.1, 95% CI 2-sided [-5.6 to 7.7]

6. Secondary Outcome: Percentage of Patients That Achieve a 15 Letter Gain in BCDVA
Description: Percentage of patients that achieve a 15 letter gain in Best Corrected Distance Visual Acuity (BCDVA) at 4 weeks, 6 weeks, 8 weeks
Time Frame: Weeks 4, week 6 and week 8
Population: LOCF, ITT population
Measure: Number; unit: percentage of subjects
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 24 | 24
percentage of subjects
  week 4 - yes | 9 | 12
  week 4 - no | 91 | 88
  week 6 - yes | 13 | 12
  week 6 - no | 87 | 88
  week 8 -yes | 13 | 17
  week 8 - no | 87 | 83
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; week 4; Test type: Superiority; p = 0.672, Chi-squared; difference in percentage = -3.8, 95% CI 2-sided [-21.3 to 13.7]
Statistical Analysis 2: Comparison: rhNGF 20 µg/ml vs Placebo; week 6; Test type: Superiority; p = 0.955, Chi-squared; difference in percentage = 0.5, 95% CI 2-sided [-18.5 to 19.6]
Statistical Analysis 3: Comparison: rhNGF 20 µg/ml vs Placebo; week 8; Test type: Superiority; p = 0.727, Chi-squared; difference in percentage = -3.6, 95% CI 2-sided [-23.9 to 16.7]

7. Secondary Outcome: Improvement in Corneal Sensitivity
Description: Improvement in corneal sensitivity was measured by the Cochet-Bonnet aesthesiometer at 4, 6 and 8 weeks.
  Corneal sensitivity is measured continuously in each patient in cm:
  * Area of the Persistent Epithelial Defect (PED) or corneal ulcer
  * All quadrants, but outside the PED or corneal ulcer area: Superior nasal, inferior nasal, superior temporal, inferior temporal.
  Improvement is defined as an increase of at least 0.5 cm in the location of concern.
Time Frame: At 4, 6 and 8 weeks after start of the treatment
Population: ITT population
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 24 | 24
cm
  week 4: number analyzed (Participants) | 20 | 17
  week 4 | 2.50 (1.821) | 1.56 (1.983)
  week 6: number analyzed (Participants) | 19 | 16
  week 6 | 2.26 (2.009) | 1.84 (2.150)
  week 8: number analyzed (Participants) | 18 | 15
  week 8 | 2.91 (2.144) | 1.83 (1.952)
  Change from baseline to week 8: number analyzed (Participants) | 18 | 15
  Change from baseline to week 8 | 1.88 (1.401) | 1.00 (1.254)
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; Test type: Superiority; p = 0.207, ANCOVA; least square mean difference = 0.6, 95% CI 2-sided [-0.4 to 1.5]

8. Secondary Outcome: Patients Experiencing Deterioration
Description: Number of patients experiencing deterioration (increase in lesion size ≥ 1mm and/or decrease in BCDVA by >5 Early Treatment Diabetic Retinopathy Study (ETDRS) letters and/or progression in lesion depth to corneal melting or perforation and/or onset of infection) in stage 2 or 3 NK from baseline to Week 8.
Time Frame: from baseline to Week 8.
Population: ITT population. As far as this endpoint is concerned, data are available (non-missing) for 18 patients out of 24 in the rhNGF group, and for 15 patients out of 24 for the vehicle group.
Measure: Number; unit: Number of subjects
Arm/Group | rhNGF 20 µg/ml | Placebo
Number analyzed (Participants) | 18 | 15
Number of subjects
  Deterioration | 0 | 2
  No deterioration | 18 | 13
Statistical Analysis 1: Comparison: rhNGF 20 µg/ml vs Placebo; Test type: Superiority; p = 0.110, Chi-squared; difference in percentage = -13.3, 95% CI 2-sided [-30.5 to 3.9]

ADVERSE EVENTS:
Time Frame: Adverse events were analyzed by study period (Controlled Treatment Period, Follow-up Period and Uncontrolled Treatment Period).
Description: The number of Participants considered in the Adverse Event Section reflects the safety subset population of the study:
  * 23 patients: rhNGF during the Controlled Treatment Period
  * 24 patients: vehicle during the Controlled Treatment Period
  * 18 patients: rhNGF during the Follow-up Period
  * 21 patients: vehicle during the Follow-up Period
  * 13 patients: vehicle during the Controlled Treatment Period and rhNGF during the Uncontrolled Treatment Period
Groups:
- rhNGF 20 µg/ml - Controlled Treatment Period; rhNGF 20 µg/ml - Follow-up Period: rhNGF 20 µg/ml eye drops solution, formulation containing anti-oxidant
  rhNGF 20µg/ml
- Vehicle - Controlled Treatment Period; Vehicle - Follow-up Period: vehicle, formulation containing anti-oxidant
  Placebo Vehicle
- Uncontrolled Treatment Period: rhNGF 20 µg/ml eye drops solution, formulation containing anti-oxidant
  Patients randomized to vehicle at baseline and not completely healed at week 8 who entered a 8-week treatment period before entering follow-up period
Arm/Group | rhNGF 20 µg/ml - Controlled Treatment Period | Vehicle - Controlled Treatment Period | rhNGF 20 µg/ml - Follow-up Period | Vehicle - Follow-up Period | Uncontrolled Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 5/18 | 2/21 | 0/13
Serious Adverse Events (participants affected / at risk) | 4/23 | 4/24 | 4/18 | 2/21 | 0/0
Other Adverse Events (participants affected / at risk) | 21/23 | 18/24 | 14/14 | 9/9 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 µg/ml - Controlled Treatment Period (N=23) | Vehicle - Controlled Treatment Period (N=24) | rhNGF 20 µg/ml - Follow-up Period (N=18) | Vehicle - Follow-up Period (N=21) | Uncontrolled Treatment Period (N=0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Corneal Thinning (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Aqueous Humour Leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Disease Progression (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | NA
decreased visual acuity (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | NA
ventral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Corneal perforation (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | NA
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Disease recurrence (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Viral gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 20 µg/ml - Controlled Treatment Period (N=23) | Vehicle - Controlled Treatment Period (N=24) | rhNGF 20 µg/ml - Follow-up Period (N=14) | Vehicle - Follow-up Period (N=9) | Uncontrolled Treatment Period (N=13)
Visual acuity reduced (Eye disorders) | 5 (5) | 5 (7) | 1 (1) | 2 (2) | 2 (2)
Eye pain (Eye disorders) | 7 (11) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Corneal Epithelium Defect (Eye disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Eye Inflammation (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Corneal Thinning (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Ocular Discomfort (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign Body Sensation In Eyes (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Posterior Capsule Opacification (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anterior Chamber Inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Deposits (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Neovascularisation (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Corneal Perforation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Discharge (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid Oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Pain (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyphaema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular Fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meibomian Gland Dysfunction (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Punctate Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative Keratitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Sensation Of Foreign Body (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Infection Intraocular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ophthalmic Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Investigations) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aqueous Humour Leakage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivochalasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Floppy eyelid syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migrane (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
LImitations and caveats non specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No